CLINICAL TRIAL: NCT06529016
Title: Using Dichoptic Therapy to Treat Intermittent Exotropia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM20027943
Record Dates: First submitted 2024-07-19; First posted 2024-07-31 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Exotropia Intermittent
Keywords: Dichoptic therapy

STUDY DESIGN:
Intervention Model Description: Prospective pilot clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Luminopia VR headset treatment (Experimental): Using Dichoptic Therapy to Improve Intermittent Exotropia Control in children ages 4-7
  Interventions: Device: Luminopia, a virtual reality headset; Other: Paper pre- survey; Other: Paper Survey

INTERVENTIONS:
Device: Luminopia, a virtual reality headset — Subjects will be provided with the equipment to use in their homes for six hours usage per week (1 hour 6 days a week), for 12 weeks.
Other: Paper pre- survey — Pre-survey to be completed by the parent and child. Questions may be skipped. Survey developed by the study team
Other: Paper Survey — Post-survey to be completed by the parent and child. Questions may be skipped. Survey developed by the study team
  Other Names: Paper post-survey

SUMMARY:
Intermittent exotropia is difficult to treat. The mainstay of treatment involves surgery, and in one long-term study authors found that as many as 60% of IXT required at least one re-operation.Patching of the non-dominant eye has also been tested in a large, multi-center randomized control trial and was not found to have a large benefit. More non-surgical treatment modalities are critical to improve the care in this condition.

DETAILED DESCRIPTION:
Luminopia, a dichoptic therapy device, was approved by the FDA in 2021 for use in amblyopia in children aged 4-7 years. The device was shown to improve vision in the amblyopic eye by lines in three months of use. Patients with strabismic amblyopia were also enrolled in the trial and found to have similar gains in vision in the amblyopic eye.

Li et al. used an investigational dichoptic therapy device in patients with intermittent exotropia and had a statistically significant improvement in ocular alignment as measured in prism diopters.The dichoptic therapy this study used is not commercially available, therefore using Luminopia to study this population may result in an immediately available non-surgical treatment for intermittent exotropia patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with IXT
* one eye that is their preferred eye
* ages 4-7
* distance control scores of <= 4

Exclusion Criteria:

* distance control scores of 5
* patients with visual acuity with vision that is worse in one eye by greater than two lines
* no preferred eye
* patients who would be unable to tolerate wearing the headset for 1 hour/day, 6 days/week, for 12 weeks.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2024-07-26 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Dichoptic therapy change of control of intermittent exotropia using the standard control score | 3 months for primary response, and 6 months after a washout period (3 months without the device)
  Improvement of the control of IXT using the Exotropia control scale that runs from 0-5. 0 meaning No exotropia noted unless dissociated, recovers in < 1 seconds (exophoria). A 5 means Constant exotropia during 30-second observation before dissociation.

SECONDARY OUTCOMES:
Change of amplitude of exotropia as measured by Alternating Prism Cover Test | 3 months for primary response, and 6 months after a washout period (3 months without the device)
  The alternate prism cover test is similar to the alternate cover test, with the addition of a prism held over one eye to quantify the misalignment. The examiner performs the alternate cover test while changing the prism over the deviated eye until the misalignment is neutralized
Change of scores from the Pediatric Eye Disease Investigator Group (PEDIG) intermittent exotropia questionnaire | 3 months for primary response, and 6 months after a washout period (3 months without the device)
  The Intermittent Exotropia Questionnaire (IXTQ) is a patient-derived, intermittent exotropia-specific instrument designed to evaluate health-related quality of life (HRQOL) in children with intermittent exotropia. The12-item assessment ivalues were converted to 0 (best) to 100 (worst)

CONTACTS AND LOCATIONS:
Overall Officials: Evan Silverstein, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States